CLINICAL TRIAL: NCT05880524
Title: Reduction of SystemiC Inflammation After Ischemic Stroke by Intravenous DNase Administration (ReSCInD)
Acronym: ReSCInD
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Collaborators: University Hospital Erlangen (Other); University Hospital Regensburg (Other)
Responsible Party: Principal Investigator, Martin Dichgans, Sponsor-Delegated Person and Principal Investigator, Ludwig-Maximilians - University of Munich
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RESCIND-1-2023; 2022-003410-37 (EudraCT Number)
Record Dates: First submitted 2023-04-30; First posted 2023-05-30 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Ischemic Stroke; Inflammatory Response
MeSH Terms: conditions — Ischemic Stroke | interventions — dornase alfa

STUDY DESIGN:
Intervention Model Description: Monocentric, randomised, placebo-controlled single-blinded, Phase 2 trial
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pulmozyme (Active Comparator): Dornase alfa; intravenous administration; 500 µg/kg
  Interventions: Drug: Dornase Alfa
- Isotonic Saline Solution (Placebo Comparator): NaCl 0,9 %; intravenous administration; 0,5 ml/kg
  Interventions: Drug: Isotonic Saline Solution

INTERVENTIONS:
Drug: Dornase Alfa — Patients will receive an intravenous dose of Dornase alfa twice within within 24±6 hours after symptom onset, administered as a bolus.
  Other Names: Pulmozyme
  Arms: Pulmozyme
Drug: Isotonic Saline Solution — Patients will receive an intravenous dose of Isotonic saline solution twice within within 24±6 hours after symptom onset, administered as a bolus.
  Other Names: NaCl 0,9%
  Arms: Isotonic Saline Solution

SUMMARY:
The goal of this (monocentric, randomised, placebo-controlled single-blinded; phase 2) clinical trial is to test the hypothesis that DNase 1 administration leads to a reduction in systemic immune response measured in patients after acute ischaemic stroke compared to control treatment.

Participants will receive intravenous DNase 1 (500 µg/kg) or placebo (NaCl 0.9%) twice within 24±6 hours after symptom onset (last seen well). Blood samples will be taken at baseline, day 1 and 3. Personal visits will occur on baseline, day 1, 3 and discharge date. A telephone interview will be conducted on day 30±3.

ELIGIBILITY:
Inclusion Criteria:

* Patients with suspected acute ischemic stroke with symptom onset (last-seen-well) until Investigational drug application of less than 12 hours.
* Consent to participate in the study.
* Age ≥ 18 years.
* NIHSS ≥10 at admission.

Exclusion Criteria:

* Presence of any of the following conditions: Sinus or cerebral venous thrombosis, intracerebral haemorrhage, subarachnoid haemorrhage on qualified imaging (cCT with CT-A or MRI with MR-A). However, petechial haemorrhagic transformations of the index infarct and cerebral microhaemorrhages may be included.
* Active malignant tumour disease in the last 6 months.
* Current known immunosuppression due to immunomodulatory medication with immunosuppressive dose or underlying immunosuppressive disease (e.g. HIV).
* Acute fulminant infectious disease in the last 7 days (fever > 38.5°C or suspected by the Investigator).
* Breastfeeding or pregnant woman, women of childbearing age without known use of contraceptives with positive urine or serum beta-human choriogonadotropin test.
* Ischemic stroke or myocardial infarction in the previous 30 days.
* Surgery in the previous 30 days, except minor dermatological or gynaecological surgery without anaesthesia and wound healing disorders and patients with thrombectomy.
* Estimated or known weight > 100 kg.
* Known allergies or intolerance to dornase alfa (Pulmozyme) or recombinant protein products derived from Chinese hamster ovary cells.
* Thrombocytopenia, leukocyte count <1500/μl.
* Known participation in another clinical trial investigating a drug and/or medical product in the last 7 days before study inclusion.
* Severe renal insufficiency with GFR≤29 ml/min/ 1.73m³ and/or renal insufficiency requiring dialysis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Concentration of interleukin-1 beta in blood of patients with acute ischemic stroke receiving Dornase alfa compared to placebo treatment with Isotonic Saline Solution. | 24±6 hours after symptom onset
  Outcome of reduced systemic immune response measured by interleukin-1 beta concentration [pg/ml] (at 24±6 hours after symptom onset) measured by Enzyme-linked Immunosorbent Assay (ELISA).

SECONDARY OUTCOMES:
cfDNA concentration in blood. | 24±6 hours after symptom onset
  Measurement of cell-free DNA (cfDNA) concentration [ng/ml] in blood at day 1 (24±6 hours after symptom onset) compared to the placebo group with experimental analysis.
DNase 1 activity in blood. | 24±6h after symptom onset
  Comparison of DNase 1 activity [µU/ml] in blood of both treatment arms measured by Enzyme-linked Immunosorbent Assay (ELISA).
Concentration of DNase 1 in blood. | 24±6h after symptom onset
  Analysis of the DNase 1 concentration [ng/ml] in patient blood treated with Dornase alfa compared to the placebo group by Enzyme-linked Immunosorbent Assay (ELISA).
Analysis of the composition of the leukocyte population in blood. | 24±6 hours after symptom onset
  Analysing the leukocyte population [%] in blood using flow cytometry in both treatment arms.
Interleukin-6 concentration in blood after treatment. | 24±6 hours after symptom onset
  Measurement of the interleukin-6 concentration [pg/ml] in blood samples (at 24±6 hours after symptom onset) measured by Enzyme-linked Immunosorbent Assay (ELISA).
Caspase 1 concentration in blood after treatment. | 24±6 hours after symptom onset
  Analysing the caspase 1 concentration [pg/ml] in blood (at 24±6 hours after symptom onset) measured by Enzyme-linked Immunosorbent Assay (ELISA).
Assessment of patient safety after Dornase alfa treatment. | 30±3 days after symptom onset
  Safety aspects of intravenous investigational drug administration in acute ischemic stroke patients will be assessed by monitoring all study patients for 30±3 days and analysis of their:
  * routine clinical diagnostics (worsening stroke is defined as a) progression, hemorrhagic transformation of the index stroke documented by radiological imaging; b) life-threatening need for intervention; c) death from the index stroke; and/or d) increasing disability (as measured by an increase of ≥ 4 points from the lowest NIHSS score measured during hospitalization, or a 1-point increase in mRS),
  * laboratory parameters (hemoglobin, platelets, neutrophil granulocytes, leukocytes, CRP, GFR, creatinine, IL-6) and
  * number of adverse events assessed by CTCAE current version.
Comparison of the incidence of infections and antibiotic treatment in both treatment arms. | 30±3 days after symptom onset
  Comparing the incidence of infections and antibiotic treatment after Dornase alfa and Isotonic Saline Solution treatment over a period of 30±3 days after symptom onset.
Functional neurological outcome scores (National Institute of Health Stroke Scale [NIHSS, 0-42] and Modified Rankin Scale [mRS, 0-6]) at both treatment arms. | 30±3 days after symptom onset
  Analysing changes of neurological scores (National Institute of Health Stroke Scale [NIHSS, 0-42] and Modified Rankin Scale [mRS, 0-6]) from baseline to last visit 30±3 days after symptom onset.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Dichgans, Prof. Dr., Study Director — Institute for Stroke and Dementia Research, LMU Hospital
Locations (1):
- Institute for Stroke and Dementia Research, Ludwig Maximilian University Munich, University Hospital, Munich, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sharma N, Dwivedi DJ, Fux L, Hayon Y, Ruderfer I, Nataf Y, Cani E, Liaw PC. Intravenous Delivery of Long-Acting Dnase I (PRX-119) In a Murine Model of Polymicrobial Abdominal Sepsis. Shock. 2026 Jan 1;65(1):76-84. doi: 10.1097/SHK.0000000000002666. Epub 2025 Jul 8. PMID 40705350
- [Derived] Di G, Vazquez-Reyes S, Diaz B, Pena-Martinez C, Garcia-Culebras A, Cuartero MI, Moraga A, Pradillo JM, Esposito E, Lo EH, Moro MA, Lizasoain I. Daytime DNase-I Administration Protects Mice From Ischemic Stroke Without Inducing Bleeding or tPA-Induced Hemorrhagic Transformation, Even With Aspirin Pretreatment. Stroke. 2025 Feb;56(2):527-532. doi: 10.1161/STROKEAHA.124.049961. Epub 2025 Jan 27. PMID 39869712